CLINICAL TRIAL: NCT05652257
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Brensocatib Following a Single Oral Administration in Healthy Male Subjects
Brief Title: A Study of the Absorption, Metabolism, and Excretion of [14C]-Brensocatib Following a Single Oral Administration in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS1007-103
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
Keywords: [14C]-brensocatib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-brensocatib (Experimental): Healthy participants will receive single oral dose of [14C]-brensocatib on Day 1 under fasted conditions.
  Interventions: Drug: [14C]-brensocatib

INTERVENTIONS:
Drug: [14C]-brensocatib — Oral solution.

SUMMARY:
The primary purpose of the study is to determine the mass balance of total radioactivity and the routes of elimination by quantifying the urinary and fecal excretion of radioactivity following a single oral administration of [14C]-brensocatib, to characterize the pharmacokinetics (PK) of brensocatib in plasma and urine, PK of total radioactivity in plasma, whole blood, urine and to determine the blood-to-plasma ratios of total radioactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index between 18.0 and 32.0 kilograms per square meter (kg/m^2), inclusive, at screening.
2. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in as assessed by the investigator (or designee).

Exclusion Criteria:

1. Positive hepatitis panel and/or positive human immunodeficiency virus test. Results consistent with previous vaccination to Hepatitis B are not exclusionary.
2. Administration of a coronavirus disease 2019 (COVID-19) vaccine in the past 14 days prior to dosing.
3. Poor peripheral venous access.
4. Have previously completed or withdrawn from this study or any other study investigating brensocatib, and have previously received brensocatib. Known allergy to brensocatib or any of the excipients used in the formulation.
5. Exposure to significant diagnostic or therapeutic radiation (e.g., serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
6. Participated in more than 3 radiolabeled drug studies in the last 12 months (previous study to be at least 4 months prior to check-in to the study site where exposures are known to the investigator or 6 months prior to check-in to the study site for a radiolabeled drug study where exposures are not known to the investigator).

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Time Curve (AUC) of Brensocatib in Plasma | Pre-dose and at multiple timepoints post-dose on Day 1 up to maximum Day 14
  Pharmacokinetics of brensocatib following a single dose in healthy participants will be assessed.
AUC∞ Plasma Brensocatib/Plasma Total Radioactivity Ratio Calculated as AUC∞ of Plasma Brensocatib Relative to AUC∞ of Plasma Total Radioactivity | Pre-dose and at multiple timepoints post-dose on Day 1 up to maximum Day 14
AUC∞ Blood/Plasma Total Radioactivity Ratio Calculated as AUC∞ of Whole Blood Total Radioactivity to AUC∞ of Plasma Total Radioactivity | Pre-dose and at multiple timepoints post-dose on Day 1 up to maximum Day 14
Amount Excreted in Urine (Aeu) of Brensocatib | Pre-dose and at multiple timepoints post-dose on Day 1 up to maximum Day 14
Total Radioactivity Expressed as Amount of [14C]-brensocatib Excreted in Urine | Pre-dose and at multiple timepoints post-dose on Day 1 up to maximum Day 14
Total Radioactivity Expressed as Amount of [14C]-brensocatib Excreted in Feces (Aef) | Pre-dose and at multiple timepoints post-dose on Day 1 up to maximum Day 14

SECONDARY OUTCOMES:
AUC of Brensocatib Metabolites in Plasma | Pre-dose and at multiple timepoints post-dose on Days 1 to 9
  Pharmacokinetics of the metabolites following a single dose of brensocatib in healthy participants will be assessed.
Number of Participants Who Experienced at Least one Adverse Event (AE) | Up to Day 14
  Safety and tolerability of a single dose of brensocatib will be determined in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No